CLINICAL TRIAL: NCT01350960
Title: A First-in-Human (FIH), Randomized, Dose-Escalation, Double-Blind, Placebo-Controlled Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SPC5001 Administered to Healthy Subjects and Subjects With Familial Hypercholesterolemia (FH)
Brief Title: Multiple Ascending Dose Study of SPC5001 in Treatment of Healthy Subjects and Subjects With FH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPC5001-901; EudraCT 2011-000489-36
Record Dates: First submitted 2011-05-05; First posted 2011-05-10 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; hyperlipidemia; LDL; HDL; PCSK9; LNA-oligonucleotide
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — SPC5001; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- saline 0.9% (Placebo Comparator)
  Interventions: Drug: Saline 0.9%
- Cohort 1 (Experimental): 0.5 mg/kg in Healthy Subjects
  Interventions: Drug: SPC5001
- Cohort 2 (Experimental): 1.5 mg/kg in Healthy subjects
  Interventions: Drug: SPC5001
- Cohort 3 (Experimental): 5.0 mg/kg in Healthy subjects
  Interventions: Drug: SPC5001
- Cohort 4 (Experimental): 10 mg/kg in Healthy subjects
  Interventions: Drug: SPC5001
- Cohort 5 (Experimental): TBD mg/kg in FH subjects
  Interventions: Drug: SPC5001

INTERVENTIONS:
Drug: SPC5001 — 3 weekly SC injections
  Arms: Cohort 1
Drug: Saline 0.9% — 3 weekly SC injections
  Arms: saline 0.9%
Drug: SPC5001 — 3 weekly SC injections
  Arms: Cohort 2
Drug: SPC5001 — 3 weekly SC injections
  Arms: Cohort 3
Drug: SPC5001 — 3 weekly SC injections
  Arms: Cohort 4
Drug: SPC5001 — 3 weekly SC injections
  Arms: Cohort 5

SUMMARY:
The purpose is to study Safety and Tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects and subjects with heterozygous Familial Hypercholesterolemia

   * Healthy male or female subjects, age 18 to 65 years, inclusive will be enrolled in Cohorts 1 through 4.
   * In Cohort 5, male or female subjects with heterozygous Familial Hypercholesterolemia, confirmed through genetic testing, without a history of cardiovascular disease (e.g. coronary artery, peripheral artery or cerebrovascular disease), hypertension or diabetes mellitus age 18-45 years, inclusive, will be enrolled.
2. BMI of 18-33 kg/m2
3. Screening hematology, clinical chemistries, coagulation and urinalysis consistent with overall good health and the following criteria are met:

   * LDL ≥.3.24 mmol/L (≥ 100 mg/dL)
   * Triglycerides (fasted) < 4.5 mmol/L (< 398 mg/dL)
   * ALT within normal limits for healthy subjects and ALT < 2 x ULN for FH subjects

Exclusion Criteria:

1. Any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential

   - History or presence of malignancy within the past year is an exclusion criterion. Subjects who have been successfully treated with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
2. Active acute or chronic infection, including, but not limited to: upper airway infection, urinary tract infection, and skin infection
3. Use of prescription medication within 14 days prior to the planned first drug administration and throughout the study. For the FH subjects statin therapy (and other lipid lowering therapies) will be prohibited within 4 weeks prior to the first study drug administration.
4. Use of non-prescription or over-the-counter medications is prohibited within 7 days prior to the planned first drug administration and throughout the study. This includes all vitamins, herbal supplements, or remedies. An exception can be made for medication or supplements that in the opinion of both the investigator and the Sponsor do not complicate or compromise the study or interfere with the study objectives.
5. Positive results on the following Screening laboratory tests: urine or serum pregnancy test (women only), alcohol breath test, urine drugs of abuse, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Regularly over 78 days
  Safety evaluation will assess adverse event (AE) profile, clinical laboratory safety tests, vital signs and ECG monitoring

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SPC5001 | up to 78 days
Lipid lowering effect | Through out the study
Area under the plasma concentration versus time curve (AUC) of SPC5001 | up to 78 days

CONTACTS AND LOCATIONS:
Overall Officials: Koos Burggraaf, MD PhD, Principal Investigator — Centre for Human Drug Research (CHDR)
Locations (1):
- Centre for Huma Drug Research (CHDR), Leiden, Netherlands

REFERENCES:
- [Derived] van Poelgeest EP, Hodges MR, Moerland M, Tessier Y, Levin AA, Persson R, Lindholm MW, Dumong Erichsen K, Orum H, Cohen AF, Burggraaf J. Antisense-mediated reduction of proprotein convertase subtilisin/kexin type 9 (PCSK9): a first-in-human randomized, placebo-controlled trial. Br J Clin Pharmacol. 2015 Dec;80(6):1350-61. doi: 10.1111/bcp.12738. Epub 2015 Oct 24. PMID 26261033